CLINICAL TRIAL: NCT04524429
Title: Quality of Life After Bariatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Adelaide (Other)
Collaborators: Central Adelaide Local Health Network Incorporated (Other Government)
Responsible Party: Principal Investigator, Antonio Barbaro, Associate Clinical Lecturer, University of Adelaide
Other Study IDs: 13441
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Bariatric Surgery Candidate; Obesity; Obesity, Morbid; Quality of Life
MeSH Terms: conditions — Obesity; Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-operative Group: This is the group of participants who suffer from obesity and are awaiting bariatric surgery.
- Post-operative Group: This is the group of participants who suffer from obesity and have received bariatric surgery.
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Procedure: Bariatric Surgery — Bariatric surgery includes sleeve gastrectomy and gastric bypass.
  Groups: Post-operative Group

SUMMARY:
This study aims to assess long term outcomes for patients who have underwent bariatric surgery. In particular, it aims to assess the quality of life of these participants.

ELIGIBILITY:
Inclusion Criteria:

* Obese, either received bariatric surgery or have been referred for bariatric surgery.

Exclusion Criteria:

* Emergency cases, Obese patients who have not been referred for bariatric surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-operative Group The pre-operative population will be patients who have been referred to TQEH bariatric clinic however have not yet had their initial appointment. The 150 participants who have been on the waiting list for the longest period of time will be included in the pre-operative group.
  Post-operative Group The post-operative population will be the 140 patients who underwent bariatric surgery at TQEH between 2008 and 2018. This resulted in 146 operations.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2020-12-20 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life before and after bariatric surgery | This represents the patients current quality of life within the last 4 weeks.
  Difference in SF-36 between post-bariatric surgical patients and representative pre-operative patients who have not undergone bariatric surgery (quality of life).

SECONDARY OUTCOMES:
Current Weight | This is the patients current weight within the last 4 weeks
  This represents the patients current weight in kilograms.
Lowest Weight | Retrospectively reviewed on average of 5 years
  This represents the patients lowest weight after bariatric surgery
Change in marker of Type 2 Diabetes Mellitus | Preoperative use compared to results within the last 4 weeks
  Using HbA1C scores and use of insulin
Change in marker of hypertension | Preoperative use compared with use in the last 4 weeks
  Number of medications used to manage condition
Change in marker of hyperlipidemia | Preoperative use compared with use in the last 4 weeks
  Number of medications used to manage condition
Change in marker of GORD | Preoperative use compared with use in the last 4 weeks
  Number of medications used to manage condition
Change in marker of OSA | Preoperative use compared with use in the last 4 weeks
  Use of CPAP

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Barbaro, MBBS, Principal Investigator — University of Adelaide, Central Adelaide Local Health Network; Matheesha Herath, MBBS, Principal Investigator — Central Adelaide Local Health Network; Raghav Goel, MBBS, Principal Investigator — Central Adelaide Local Health Network; Gayatri Asokan, MBBS, FRACS, Principal Investigator — Central Adelaide Local Health Network; Markus Trochsler, MD, FMH, MMIS, FRACS, Study Director — Central Adelaide Local Health Network; Harsh Kanhere, MS, FRACS, AFRACMA, Study Director — Central Adelaide Local Health Network
Locations (1):
- The Queen Elizabeth Hospital, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No